CLINICAL TRIAL: NCT00903552
Title: A Phase 2a Randomized, Double Blind, Placebo Controlled Trial to Evaluate the Safety and Immunogenicity of a Trivalent Seasonal Influenza Virus-Like Particle (VLP) Vaccine (Recombinant) in Healthy Adults
Brief Title: Trial to Evaluate Safety and Immunogenicity of Trivalent Seasonal Influenza Virus-Like Particle (VLP) Vaccine (Recombinant)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NVX 755.203
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Seasonal Influenza

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose (Experimental)
  Interventions: Biological: Influenza VLP Vaccine
- PBS (Placebo Comparator)
  Interventions: Biological: Placebo
- High Dose (Experimental)
  Interventions: Biological: Influenza VLP Vaccine

INTERVENTIONS:
Biological: Influenza VLP Vaccine
  Arms: High Dose; Low Dose
Biological: Placebo — phosphate-buffered saline (PBS)
  Arms: PBS

SUMMARY:
This is a phase 2A randomized, double blind, placebo controlled trial to evaluate the safety and immunogenicity of a trivalent seasonal influenza virus-like particle (VLP) vaccine (recombinant) in healthy adults.

DETAILED DESCRIPTION:
The primary study objectives are:

* To assess the tolerability and safety of the Influenza VLP Vaccine
* To assess the immunogenicity of the Influenza VLP Vaccine as measured by hemagglutination inhibition (HAI) antibody titers to each of the component viral strains

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female 18 to 49 years of age at the time of the vaccination
2. Informed consent must be obtained from the subject prior to beginning any study specific procedures indicating that they understand the purpose of this study and are willing to adhere to the procedures described in this protocol
3. Available by telephone (Novavax, Inc. CONFIDENTIAL 22 Apr2009; NVX 755.203 Version 2.0 Page 22 of 52)
4. Free of obvious health problems or chronic illnesses (i.e., recent exacerbation or acute episode of chronic illness in the last 6 months) as established by medical history, review of systems, and clinical examination before entering the study:

   * This includes any mental condition that would interfere with subject self-assessment
   * Subjects with a pre-existing chronic disease (such as but not limited to hypertension, diabetes, hypothyroidism) will be allowed to participate if the disease is stable (stable disease is defined as no new onset of exacerbation of pre-existing chronic disease 6 months prior to study vaccine injection)
5. If subject is of childbearing potential, she must be abstinent or have used adequate contraceptive precautions (e.g., intrauterine contraceptive device; oral contraceptives or other equivalent hormonal contraception) for 2 months prior to vaccination. She must also have a negative pregnancy test at study entry and must agree to continue such precautions for three months after vaccination

Exclusion Criteria:

1. Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the administration of the study vaccine, or planned use during the study period
2. Has received any other licensed or investigational influenza vaccine within 12 months prior to enrollment in this study or expected receipt of any influenza vaccination before the final immune response blood collection
3. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the administration of the study vaccine

   * The use of inhaled and nasal steroids will be permitted
4. Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination
5. Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or during the study
6. Acute disease at the time of enrollment. Acute disease is defined as the presence of a moderate or severe illness with or without fever > 100.5°F
7. Acute clinically significant pulmonary (e.g., asthma), cardiovascular, hepatic or renal functional abnormality as determined by physical examination or laboratory screening tests
8. Major congenital defects
9. History of any neurological disorders or seizures, with the exception of febrile seizures during childhood
10. Pregnant or lactating female
11. Females planning to become pregnant or planning to discontinue contraceptive precautions within 60 days of enrollment in this study
12. Any condition that in the opinion of the investigator would interfere with evaluation of the vaccine or interpretation of study results

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To assess the tolerability and safety of the Influenza VLP Vaccine | 10 days, 6 months
The Influenza VLP Vaccine will be immunogenic | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Thomas, Ph.D., Study Director — Novavax, Inc.
Locations (2):
- United States (2):
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - SNBL Clinical Pharmacology Center, Baltimore, Maryland